CLINICAL TRIAL: NCT05491850
Title: Effects of Moderate Physical Activity on Early Symptoms of Peripheral Diabetic Neuropathy in Type-II Diabetes: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Waqar Ahmed Awan, Principal Investigator, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIPHAH/FR&AHS/Letter-0985
Record Dates: First submitted 2022-07-31; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Peripheral Diabetic Neuropathy
Keywords: Type 2 diabetes mellitus, moderate physical activity, HbA1c, diabetic neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Physical Activity Group (Experimental): The Experimental Group gets moderate physical activity. Elliptical will be performed at least 5 days/per week. Moderate intensity, corresponding approximately to 40-60% of Vo2max (maximal aerobic capacity) 150 min/week of exercise undertaken at moderate intensity or greater. Warm-up and Dynamic stretching is given before and static stretching is given after moderate physical activity.
  Interventions: Other: Moderate Physical Activity for Peripheral Diabetic Neuropathy
- Non Specific Physical Activity Group (No Intervention): The Control group continues their regular medication for diabetic neuropathy.

INTERVENTIONS:
Other: Moderate Physical Activity for Peripheral Diabetic Neuropathy — Moderate physical activity can increase movement and heart rate are particularly important for people suffering with peripheral neuropathy. Physical activity can improve blood circulation, which strengthens nerve tissues by increasing the flow of oxygen.
  Arms: Moderate Physical Activity Group

SUMMARY:
This study determines the effects of moderate physical activity on early symptoms of peripheral diabetic neuropathy in type-II diabetes. Most of the literature shows the impact of physical activity to manage/controlling diabetes. Some studies were conducted on animals to study the impact of physical activity on diabetic neuropathy and neurogenesis. There is no study on the impact of physical activity to manage early symptoms of peripheral diabetic neuropathy in patients with type-II diabetes in humans. This study finds the impact of moderate physical activity to manage early symptoms of peripheral diabetic neuropathy in patients with type-II diabetes in humans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type-II Diabetes
* Diagnosed cases of Peripheral Diabetic Neuropathy
* Peripheral Diabetic Neuropathy Stage 1 & 2
* Numbness or reduced ability to feel pain or temperature changes.
* Tingling or burning sensation.
* Sharp pains or cramps.
* Increased sensitivity to touch
* Males and females
* Age: 35-65
* HbA1c above 6.5
* Mild activity level on IPAQ-7 (< 150min/per week)
* Berg Balance Scale score (< 45)

Exclusion Criteria:

* Cardiac Issues
* Any neurological issue
* Lower limb deformity
* Acute injury
* Hip and Knee OA
* Patients with walking difficulty
* Diabetic foot

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Effect of moderate physical activity on early symptoms of peripheral diabetic neuropathy in type-II diabetes | 2 Months
  Research Hypothesis

CONTACTS AND LOCATIONS:
Locations (1):
- RHS Rehabilitation Center, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No